# Examining Variables Affecting Patient Participation in Clinical Trials for Tinnitus: Investigating Tinnitus Clinical Trials

Informed Consent Form for Participation in <a href="Power Clinical Trial's">Power Clinical Trial's</a>
Observational Study

Date: March 30, 2023

Welcome to Our Observational Clinical Study: An Introduction

Thank you for considering participation in our research project. We understand that you may have questions and concerns, which is why we want to ensure that you have all the necessary information before making a decision. Your consent is required for participation, but you are under no obligation to do so and may withdraw at any time.

This brief summary provides an overview of the study, but we encourage you to review the more detailed information in the consent form. The primary procedures of this observational clinical study involve completing questionnaires and follow-up calls to understand why patients choose to enroll, remain, or withdraw from clinical trials. These procedures have been designed to minimize any risks to participants, and as an observational study, there may not be any direct medical benefits.

However, the data collected can be used to identify ways to improve clinical trial participation rates and ultimately benefit patients with tinnitus. By participating in this study, you have the opportunity to contribute to the advancement of medical research and the improvement of clinical trial practices.

The findings of this study will provide valuable insights into the factors affecting clinical trial participation rates. This information can be used to improve recruitment strategies and patient engagement in clinical trials, ultimately benefiting tinnitus patients. However,

we want to emphasize that participation is voluntary and declining to participate will not affect your rights or privileges.

We want to ensure that you are fully informed before making a decision about participation. We encourage you to review the consent form carefully and ask any questions you may have. It is recommended that you discuss the study with your family, friends, trusted advisors, and healthcare professionals to make an informed decision. Remember that your participation is entirely voluntary, and you have the right to withdraw at any time without consequences.

#### The Importance of This Clinical Trial

Clinical trials are essential in finding new and improved treatments for tinnitus, but it is crucial that the participation rates of these trials accurately represent the larger population. This clinical trial aims to understand the various factors that affect a patient's decision to enroll, discontinue, or resume participation in a tinnitus clinical trial.

Our objective is to increase clinical trial participation rates by identifying and understanding the reasons for underrepresented groups' low participation rates. We believe that by identifying these factors, we can develop better strategies to increase participation rates in future clinical trials.

We recognize that participating in this clinical trial is entirely voluntary, and participants have the right to withdraw at any time without any consequences. The study's primary procedures involve answering questionnaires and making follow-up calls, with minimal risk to the participants. We encourage potential participants to review the consent form carefully and discuss it with their families, friends, trusted advisors, and healthcare professionals before making a decision.

#### Clinical Trial Process

We are conducting an observational clinical research study to understand why tinnitus patients enroll, withdraw, or complete clinical trials. As a participant in an interventional trial, you have been invited to take part in this study. Our research team will use electronic medical record systems to identify potential participants who meet our study's criteria. If you choose to participate, our staff will provide you with a consent form to sign, and they will explain the study's objectives and your rights as a participant.

The study will involve completing a questionnaire every two weeks and participating in phone or video interviews with our research team every three months. These questionnaires and interviews will ask about your demographics, medical history, and reasons for enrolling, withdrawing, or completing the clinical trial. All information will be kept confidential, and you will be assigned a unique identifier instead of using your name.

The data collected will be analyzed using statistical methods to identify the factors that influence patient participation in clinical trials. The results of this study will be used to improve the recruitment and retention of tinnitus patients in future clinical studies. It is important to note that participation in this study is voluntary, and you have the right to withdraw at any time without consequence.

### Can Clinical Study Benefit You?

Participating in an observational clinical research study for tinnitus may not directly benefit participants since it does not involve experimental therapies. However, patients with tinnitus can contribute to medical research that can lead to improved treatment options in the future.

Moreover, participants may receive expert care and attention during the study. Nevertheless, it is essential to consider the potential advantages and drawbacks of participation based on each individual's unique circumstances and goals. Patients are encouraged to discuss their options with their healthcare provider and the study team before making a decision.

# Stopping the Clinical Trial

Participants in clinical studies should be aware that there are several reasons why their participation may be stopped, even if they do not agree with the decision. These reasons could be due to external factors such as the study being suspended or terminated, the withdrawal, suspension or removal of funding, or the study no longer being considered in the best interests of the participants.

There are also participant-related reasons why the researchers or sponsor may decide to discontinue involvement in the study. For example, if the participant's health deteriorates during the course of the study, or if they become pregnant, their participation may be stopped. If the participant decides not to proceed with the research

after being informed of any changes that may affect them, or if they fail to follow the study's protocols, their involvement may also be terminated.

It is important for participants to understand that stopping their involvement in the study does not necessarily mean they are no longer eligible for medical treatment or care. The study team will work with the participant and their healthcare provider to ensure that they receive appropriate follow-up care.

#### Our Clinical Trial Versus Other Tinnitus Clinical Trials

As a patient considering participating in a tinnitus clinical trial, it's important to understand the differences between these trials and other clinical trials. Tinnitus clinical trials may involve different types of interventions, such as chemotherapy, radiation therapy, or surgical procedures, depending on the specific trial's goals. These interventions can have various risks and benefits, which will be explained in detail in the informed consent form. It's essential to carefully read and understand this document before deciding whether to participate.

Furthermore, unlike other clinical trials, <u>tinnitus trials</u> may have unique eligibility criteria that may exclude certain patients based on factors such as age, illness stage, or care regimes. It's essential to discuss these criteria with your doctor and the study team to determine whether you meet the trial's requirements.

For more information on the different tinnitus studies, you can go to clinicaltrial.gov and search for the specific condition and filter according to your location so that you can see a list of studies involving tinnitus patients. You can also check Power's reference site if you are looking for active tinnitus clinical trials looking for participants.

# More Reads on Clinical Trial Representation

For those looking to expand their knowledge on the topic of clinical trial diversity, there are numerous online resources available. Below are a few articles that may be of interest to you:

Rochon, Paula A., Philip B. Berger, and Michael Gordon. "The evolution of clinical trials: inclusion and representation." *Cmaj* 159, no. 11 (1998): 1373-1374.

Rochon, Paula A., Philip B. Berger, and Michael Gordon. "The evolution of clinical trials: inclusion and representation." *Cmaj* 159, no. 11 (1998): 1373-1374.

# Participant's Consent

When you sign this consent agreement, you are indicating your understanding and acceptance of the terms and conditions outlined below:

Firstly, you have thoroughly read and comprehended the informed consent form, and before making your decision to participate, you are encouraged to discuss the information provided with others and seek alternative perspectives.

Secondly, you have received satisfactory answers to all of your queries and concerns about the research project and its methods, as well as all the information necessary to participate in the study.

Thirdly, you have considered the benefits, risks, and other alternatives to participating in the research, and are participating voluntarily without any coercion.

Fourthly, your decision to participate or not will not affect your ability to exercise your legal rights, and you can withdraw your participation from the study at any time without any negative consequences.

Lastly, if there are any significant updates or changes made to the research study that may affect your decision to continue participating, you will be informed immediately.

| Participant's Signature | | |
|-------------------------|--------------------------|------|
| Name of Participant | Signature of Participant | Date |

| Statement of | f Research | her Getting | Consent: |
|--------------|------------|-------------|----------|

As the researcher getting the consent for this study, I confirm that I have provided the patient with a thorough explanation of the research and have addressed any concerns or inquiries they had. Additionally, I have confirmed that the patient's decision to participate is completely voluntary and based on their full understanding of the information provided.

| Signature of the Research | her Who Obtained the Con | sent |
|---------------------------|--------------------------|------|
| Name of Researcher | Signature of Researcher | Date |